CLINICAL TRIAL: NCT04286217
Title: Study Using OCT_SD to Diagnose Impending Hypertensive Emergency: Relationship to Clinical Findings, Imaging and Outcomes
Brief Title: SD-OCT Measurement of the Human Retina in Pregnancy With Pre-existing or De Novo Hypertension and Without Hypertension
Status: Active, not recruiting | Type: Observational
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Other Study IDs: REB15-0374
Record Dates: First submitted 2020-01-07; First posted 2020-02-26 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-01

CONDITIONS: Pregnancy Induced Hypertension; Pregnancy Related
Keywords: human pregnancy; hemodynamic changes in pregnancy; macular thickness; microcirculation; autoregulation; spectral domain optical coherence tomography
MeSH Terms: conditions — Hypertension, Pregnancy-Induced

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (14):
- No prior hypertension (HTN); no HDP in pregnancy: No pre-existing hypertension, incident pregnancy not complicated by a hypertensive event
- No prior HTN; de novo HDP, GH type; no macular injury: No pre-existing hypertension, incident pregnancy complicated by new onset gestational hypertension, but no abnormal SD-OCT findings in the eye
- No prior HTN; de novo HDP, GH type; macular injury found: No pre-existing hypertension, incident pregnancy complicated by new onset gestational hypertension, with abnormal SD-OCT findings in the eye consistent with possible hyperperfusion injury
- No prior HTN; de novo HDP, PE type; no macular injury: No pre-existing hypertension, incident pregnancy complicated by new onset preeclampsia, but no abnormal SD-OCT findings in the eye
- No prior HTN; de novo HDP, PE type; macular injury found: No pre-existing hypertension, incident pregnancy complicated by new onset preeclampsia, with abnormal SD-OCT findings in the eye consistent with possible hyperperfusion injury
- No prior HTN; no HDP in pregnancy; postpartum HDP: No pre-existing hypertension, incident pregnancy not complicated by a hypertensive event, patient developed postpartum HDP, either gestational hypertension or preeclampsia, with abnormal SD-OCT findings in the eye consistent with possible hyperperfusion injury
- Pre-existing HTN; no HDP in pregnancy: Pre-existing hypertension, incident pregnancy not complicated by a hypertensive event
- Pre-existing HTN; de novo HDP, GH type; no macular injury: Pre-existing hypertension, incident pregnancy complicated by new onset gestational hypertension, but no abnormal SD-OCT findings in the eye
- Pre-existing HTN; de novo HDP, GH type; macular injury found: Pre-existing hypertension, incident pregnancy complicated by new onset gestational hypertension, with abnormal SD-OCT findings in the eye consistent with possible hyperperfusion injury
- Pre-existing HTN; de novo HDP, PE type; no macular injury: Pre-existing hypertension, incident pregnancy complicated by new onset preeclampsia, but no abnormal SD-OCT findings in the eye
- Pre-existing HTN; de novo HDP, PE type; macular injury found: Pre-existing hypertension, incident pregnancy complicated by new onset preeclampsia, with abnormal SD-OCT findings in the eye consistent with possible hyperperfusion injury
- Pre-existing HTN; no HDP in pregnancy; postpartum HDP: Pre-existing hypertension, incident pregnancy not complicated by a hypertensive event, patient developed postpartum HDP, either gestational hypertension or preeclampsia,with abnormal SD-OCT findings in the eye consistent with possible hyperperfusion injury
- Other causes of macular injury leading to HDP: Other causes of abnormal SD-OCT findings in the eye consistent with possible hyperperfusion injury leading to HDP, either gestational hypertension or preeclampsia
- Other causes of macular injury not leading to HDP: Other causes of abnormal SD-OCT findings in the eye consistent with possible hyperperfusion injury not leading to HDP

SUMMARY:
The complications of long-standing severe and acute severe elevations in systemic blood pressure (hypertension) may involve large vessels as well as smaller vessels, these latter comprising what is known as the microcirculation. Diseases of the microcirculation include stroke, dementia, and end stage renal disease to name a few. The microcirculation of the brain (and kidneys) possess a reflex called autoregulation that protects the downstream organ from fluctuations in blood pressure and blood flow. The neurosensory retina of the eye is a forward extension of brain and has a similar microcirculation to that of brain, including the presence of blood retinal barriers and the ability to autoregulate. One of the consequences of very severe hypertension is breakthrough of the autoregulatory reflex with hyperperfusion injury and edema formation. Currently, physicians and scientists have no tools to visualize or measure the human microcirculation or the autoregulatory reflex. SD-OCT is an advanced imaging technology that has a spatial resolution 1000-10,000 times greater than CT or MRI. It is the standard of care for identification and follow-up of structural diseases of the eye. The question this research proposal attempts to answer is whether SD-OCT is able to detect edema or other evidence of structural damage in the eyes in patients in the midst of, or following an episode of very severe hypertension. Pregnant women were chosen to be the focus of this study because: 1) pregnant women are generally young and would be expected to possess a normal microcirculation, 2) the occurrence of new-onset hypertension in pregnancy is high, occurring in 5-10% of all pregnancies, 3) there are established prediction rules that allow one to select and compare women at high- or low-risk of developing hypertension in pregnancy, and finally 4) the spectrum of hypertensive injury in pregnancy ranges from minor elevations in systemic blood pressures to eclampsia, the most severe, life-threatening form of hypertensive injury possible. All this is occurs within a 9-month time window defining human pregnancy. Thus, the investigators are proposing to examine the eyes of women using SD-OCT at low- and high-risk of developing hypertension in pregnancy to determine if, when and how this injury is occurring and its relationship to blood pressures.

DETAILED DESCRIPTION:
This is a prospective observational cohort study that was undertaken at Foothills Medical Centre, University of Calgary, Calgary, Canada. Recruitment began in October 2013 and clinical follow-ups completed in May 2017.

Data was collected at enrolment (< 20 weeks gestation), at every follow-up clinical encounter with the Foothills Hospital High-risk Obstetrical clinic between 20 weeks gestation and delivery, at delivery itself, and at least 1 additional encounter in the non-pregnant state, usually postpartum. Demographic information including participant age, gestational age, medical co-morbidities, medications, clinical symptoms, weight, height, automated office blood pressure and all investigations ordered by managing physicians were recorded. In addition, macular thickness was measured at each encounter using spectral domain optical coherence tomography (SD-OCT). Obstetrical and neonatal outcomes were collected from standardized birth and delivery records.

SD-OCT images were performed by a trained physician or research assistant according to the following standardized technique. The same Zeiss Cirrus 4000 SD-OCT instrument was used for all retinal images. Two SD-OCT images were obtained from each eye at each clinical encounter without dilation of the pupil at a scanning resolution of 512 A-scans x 128 B-scans over a 6 mm square grid focused on the fovea. Between sequential sessional measurements (i.e., right eye first measurement, right eye second measurement, etc.) participants were instructed to remove their face from the examining platform and the instrument was reset to default parameters in order to match the effect of an independent scan. Scans were examined systematically for signal strength, definition of the vessel architecture, centrality and motion artifact to determine image quality, and the better of the 2 images was prospectively selected for analysis. Macular thickness was measured from the internal limiting membrane to the retinal pigment epithelium, a standard method completed by the instrument on every retinal scan. All scans were referenced to the image obtained from the same individual in the non-pregnant state to determine interval change over the pregnancy.

Given the exploratory nature of this study and its small subject numbers, the research team considered both standard summary statistics and measures of individual response. In respect to the latter, a decision support tool was derived before starting the study whereby 'clinically meaningful change' was arbitrarily defined as a directionally identical difference ≥ ±4 µm (the test re-test coefficient of repeatability of the instrument) in 3 or more contiguous segments on the Early Treatment of Diabetic Retinopathy Study (ETDRS) grid [1] in a single eye. This summary measure was subsequently tested against the frequency of appearance of all possible combinations of ETDRS segments possessing that and other levels of differential change in a null difference distribution comprised of 1370 paired images collected on all participants enrolled in SD-OCT studies managed by the PI as of May 2017. This tool identifies a statistically significant interval change compared to the expected null difference at a P-value = 0.046. Assessment of this parameter is ongoing and will be published separately.

Participant characteristics were summarized by descriptive statistics using means and standard deviation (SD) for continuous variables and frequencies for categorical variables. A 95% confidence interval (95%CI) was computed for each outcome parameter. Statistical significance was defined as a P-value <0.05. A linear mixed-effects model was used to estimate macular thickness at the 3 gestational intervals with random effects considered at three hierarchical levels: patient level, eye side (right or left) and position on the ETDRS grid. A continuous autocorrelation structure was used to adjust for correlation of variables repeatedly measured at differing clinical encounters.

ELIGIBILITY:
Inclusion Criteria:

Cohort I Women at Low-risk for Developing an HDP (possessing none of the high risk variables outlined in Cohort II below)

Cohort II Women at High-risk for Developing an HDP

* chronic hypertension
* prior preeclampsia
* prior gestational hypertension
* chronic kidney disease, or
* ≥ 2 of the following: age >35 years, body mass index (BMI) > 30 kg/m2, twin or multiple gestation pregnancy, non-Caucasian ethnicity

Exclusion Criteria:

* pre-existing type 1 or type 2 diabetes mellitus
* vasculitis
* known or observed retinal disease at enrolment

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women aged 18-45 years and at < 20 weeks gestation will be recruited from an outpatient obstetrical internal medicine clinic at the Foothills Medical Centre in Calgary, Canada into 2 cohorts depending upon their risk for developing a hypertensive disorder of pregnancy (HDP).
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2013-10-30 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
SD-OCT measured change in retinal macular thickness during pregnancy at each gestational period for all study subgroups | At < 20 weeks gestation, from 20 weeks gestation up to before delivery, and at delivery
  The observed change in retinal macular thickness at each gestational period referenced to its baseline measurement in the non-pregnant state will be characterized using both our clinical decision support tool and summary statistics and comparisons made between each subgroup in the study. Some subgroups such as those examining pre-existing and do novo hypertension, or those looking separately at gestational hypertension and preeclampsia may be combined if the pattern of end-tissue response of the retina is the same.

SECONDARY OUTCOMES:
Relationship of mean arterial blood pressure to observed macular response in pregnancy at each gestational interval for all study subgroups | At < 20 weeks gestation, from 20 weeks gestation up to before delivery, and at delivery
  An anticipated relationship between mean arterial blood pressure and macular response (change in macular thickness brought about by hemodynamic factors, including a 1.5-fold increase in cardiac output that is known to peak between 16 and 20 weeks gestation [2], and a 1.3-1.4-fold increase in circulating blood volume peaking in late pregnancy [3]) will be examined by regression analysis. Also, mean arterial pressures will be averaged over each gestational interval for each individual, and summary statistics will be compiled and compared for those in each subgroup. Finally, if hyperperfusion injury is observed to occur in the retina in pregnancy, mean arterial pressure, symptoms/clinical findings, and laboratory abnormalities at the time where macular injury is first detected will be noted and compared for accuracy in defining that event.

OTHER OUTCOMES:
Relationship of breach of microcirculatory autoregulatory integrity of the eye, if observed, to breach in other regional circulations | At < 20 weeks gestation, from 20 weeks gestation up to before delivery, and at delivery
  Examples, the kidney where findings of new onset and worsening proteinuria, or elevation of liver enzymes presumably due to gut/visceral edema would be an important outcome of interest in this study. All findings noted and comparisons made, as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Herman, MD, Principal Investigator — University of Calgary

IPD SHARING:
Plan to Share IPD: No
There is no plan at this time.

REFERENCES:
- [Background] Huang J, Liu X, Wu Z, Xiao H, Dustin L, Sadda S. Macular thickness measurements in normal eyes with time-domain and Fourier-domain optical coherence tomography. Retina. 2009 Jul-Aug;29(7):980-7. doi: 10.1097/IAE.0b013e3181a2c1a7. PMID 19584656
- [Background] Conti E, Zezza L, Ralli E, Caserta D, Musumeci MB, Moscarini M, Autore C, Volpe M. Growth factors in preeclampsia: a vascular disease model. A failed vasodilation and angiogenic challenge from pregnancy onwards? Cytokine Growth Factor Rev. 2013 Oct;24(5):411-25. doi: 10.1016/j.cytogfr.2013.05.008. Epub 2013 Jun 22. PMID 23800655
- [Background] Kanasaki K, Kalluri R. The biology of preeclampsia. Kidney Int. 2009 Oct;76(8):831-7. doi: 10.1038/ki.2009.284. Epub 2009 Aug 5. PMID 19657323
- [Background] Magee LA, Pels A, Helewa M, Rey E, von Dadelszen P; Canadian Hypertensive Disorders of Pregnancy Working Group. Diagnosis, evaluation, and management of the hypertensive disorders of pregnancy: executive summary. J Obstet Gynaecol Can. 2014 May;36(5):416-41. doi: 10.1016/s1701-2163(15)30588-0. English, French. PMID 24927294
- [Background] Wolf M, Shah A, Jimenez-Kimble R, Sauk J, Ecker JL, Thadhani R. Differential risk of hypertensive disorders of pregnancy among Hispanic women. J Am Soc Nephrol. 2004 May;15(5):1330-8. doi: 10.1097/01.asn.0000125615.35046.59. PMID 15100374